CLINICAL TRIAL: NCT02061722
Title: [PETDE10] Imaging of Phosphodiesterase 10 A (PDE10A) Enzyme Levels in the Living Human Brain of Huntington´s Disease Gene Expansion Carriers and Healthy Controls With Positron Emission Tomography
Brief Title: [PETDE10] Imaging of PDE10A Enzyme Levels in Huntington's Disease Gene Expansion Carriers and Healthy Controls With PET.
Acronym: PEARL-HD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CHDI Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHDIKI1201/PET-HD-PDE10A
Record Dates: First submitted 2014-02-03; First posted 2014-02-13 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-03

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — Magnetic Resonance Spectroscopy; 2-(2-(3-(4-(2-fluoroethoxy)phenyl)-7-methyl-4-oxo-3,4-dihydroquinazolin-2-yl)ethyl)-4-isopropoxyisoindoline-1,3-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET Imaging with [18F]MNI-659 (Experimental): All subjects (both HDGECs and HCs) will receive single intravenous doses of the radioligands [11C]raclopride (non-investigational medicinal product [NIMP]) and [18F]MNI-659 (investigational medicinal product [IMP]).
  The radioligands [11C]raclopride and [18F]MNI-659 will be administered at doses less than 10 micrograms, i.e. within the micro dosing concept, and no pharmacological effects are expected.
  The injected radioactivity of [11C]raclopride will be 300 MBq/70 kg of body weight ± 10%.
  The injected radioactivity of [18F]MNI-659 will be 185 MBq/70 kg of body weight ± 10%.
  Interventions: Radiation: PET Imaging with [18F]MNI-659

INTERVENTIONS:
Radiation: PET Imaging with [18F]MNI-659 — The radioligands [11C]raclopride and [18F]MNI-659 will be administered at doses less than 10 micrograms, i.e. within the micro dosing concept, and no pharmacological effects are expected.
  The injected radioactivity of [11C]raclopride will be 300 MBq/70 kg of body weight ± 10%.
  The injected radioactivity of [18F]MNI-659 will be 185 MBq/70 kg of body weight ± 10%.

SUMMARY:
The aim of this study is to measure the availability of the PDE10A enzyme in Huntington disease gene expansion carriers (HDGECs) using the recently developed radioligand [18F]MNI-659. The study will be cross-sectional, examining HDGECs at different stages of the disease (pre-manifest, stage 1 and stage 2), in comparison with Healthy Controls (HCs). The HDGECs included in this study will be recruited from the large database of the REGISTRY (NCT01590589) or ENROLL-HD (NCT01574053) studies.

DETAILED DESCRIPTION:
The study will be organized in an "adaptive-like" mode. Initially a cohort of 5 HDGECs and 5 HCs will be studied. The data obtained in the first cohort will be analysed and depending on the variability of the data, there will be approximately 10 HDGECs and an equal number of HCs in the second cohort and the size of the third cohort may be altered to in total include approximately 45 HDGECs and an equal number of HCs.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to give full informed consent in writing, and have read and signed the informed consent
* Age 18 to 70 years, inclusive
* HCs: Healthy according to medical history, physical examination, ECG, vital signs, laboratory assessment and MRI, with a body mass index between 19 and 27 (both inclusive)
* HDGECs: Otherwise healthy according to medical history, no co-morbidity of psychotic disorders, physical examination, vital signs and laboratory assessments
* HDGECs:

(A) HD Stage 1 or HD Stage 2: Patients with a clinical diagnosis of HD, defined by the presence of noticeable motor disorder and 40 CAG repeats (HD stage 1: Total Functional Capacity (TFC) 11-13, HD stage 2: TFC 7-10); (B) Pre-manifest: Subjects that are carriers of the mutant Huntingtin gene with ≥40 CAG repeats, a disease burden score ≥ 275 (calculated by the equation ((CAGn-35.5) X age)), and a Total Motor Score (TMS) ≤ 5.

* Able and willing to travel to Stockholm
* Willing to comply with use of adequate contraceptive measures:

Exclusion Criteria:

* Any disease, condition or concomitant medications that significantly compromises the function of the body systems and that, in the opinion of the Investigator might interfere with the conduct of the study or the interpretation
* Regular use of any medication prohibited by this protocol with the exception for Viagra, Levitra and Cialis, which may be temporarily discontinued prior to the PET measurements
* HDGECs: History of other neurological condition (including brain surgery, intracranial haematoma, stroke/cerebrovascular disorders, epilepsy), co-morbidity of psychotic disorders
* HCs: Anamnesis/medical history of neurological conditions (Alzheimer´s disease, dementia, Parkinson´s disease, brain surgery, intracranial haematoma, stroke/cerebrovascular disorders, epilepsy) or psychiatric conditions schizophrenia, depression, bipolar disorder, attention-deficit hyperactivity disorder)
* HCs: Family history of HD
* History of or current alcohol or drug abuse or dependence
* History of anaphylactoid or anaphylactic reactions to any allergen including drugs and contrast media
* Haematological or biochemical parameters that are outside the normal range and are considered clinically significant by the Investigator
* Clinical relevant findings in the 12-lead ECG as determined by the evaluating physician
* Donation of blood (450 mL) within three months prior to Visit 3
* Contraindication to MRI, such as known claustrophobia, presence of metal devises or implants (e.g. pacemaker, vascular- or heart- valves, stents, clips), metal deposited in the body (e.g. bullets or shells), or metal grains in the eyes
* Participating in a clinical trial within the past 3 months
* HCs: previous participation in another PET study
* Positive viral test result for Hepatitis B or C or HIV 1 or 2
* Female subjects: breast-feeding or positive pregnancy test at screening or at Visit 3
* Contraindication for arterial cannulation (by assessment of Allen's test)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the distribution volume (VT) in the striatum (caudate and putamen), globus pallidus, and ventral striatum estimated using kinetic and graphical analysis. Thalamus, cortex and cerebellum will also be examined. | Visit 3: For HD subjects, this will occur within 90 days from the Screening Visit. For Healthy Controls, this will occur within 28 days of Screening visit.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Landwehrmeyer, MD, PhD, Principal Investigator — Ulm University Hospital; Cristina Sampaio, MD, PhD, Study Director — CHDI Foundation, Inc.
Locations (8):
- The Memory Clinic, Rigshopitalet, Copenhagen, Denmark
- Leiden University Medical Center, Department of Neurology, Leiden, Netherlands
- University of Oslo, Nevrologisk poliklinikk, Oslo, Norway
- Sweden (5):
  - Skane Universitetssjukhus Lund, Neurologiska kliniken, Lund
  - Karolinska Universitetssjukhus, Huddinge, Stockholm
  - Karolinska University Hospital, Stockholm
  - KTA Karolinska Trial Alliance, Stockholm
  - Neurologkliniken Akademiska sjukhuset, ing 85, Uppsala